# Dashboard Activated Services and tele-Health for Heart Failure (DASH-HF) Study

# **Study Protocol**

**Principal Investigator:** Boback Ziaeian, MD, PhD, FACC, FAHA

Assistant Professor of Medicine

David Geffen School of Medicine at UCLA VA Greater Los Angeles Healthcare System

**Trial Statistician:** Boback Ziaeian, MD, PhD, FACC, FAHA

**Protocol Authors:** Aradhana Verma, MD

Boback Ziaeian, MD PhD

SAP Version: 1.0

NCT Number: Not assigned

**Date:** 7/20/21

# **Table of Contents**

| Abbr | eviations and Definitions | 3 |
|---|---|---|
| Intro | duction | 4 |
| Study | or Objectives | 5 |
| Study | / Methods | 7 |
| 4.1 | General Study Design and Plan | |
| 4.2 | Inclusion-Exclusion Criteria and General Study Population | |
| 4.3 | Randomization and Blinding | |
| Safet | у | |
| Adve | rse Events | |
| Refer | rences | 15 |
| Listing of Tables, Listings, and Figures | | |
| Supp | lemental Materials | 17 |
| | Study<br>Study<br>4.1<br>4.2<br>4.3<br>Safet<br>Adve<br>Refer<br>Listin | <ul> <li>4.2 Inclusion-Exclusion Criteria and General Study Population</li> <li>4.3 Randomization and Blinding</li> <li>Safety</li> <li>Adverse Events</li> <li>References</li> </ul> |

# 1 Abbreviations and Definitions

ACE angiotensin-converting enzyme inhibitor
ADHFD Academic Detailing Heart Failure Dashboard

AKI acute kidney injury

ARB angiotensin II receptor blockers

ARNI angiotensin receptor neprilysin inhibitor

HF heart failure

HFrEF heart failure with reduced ejection fraction

LVEF left ventricular ejection fraction

MRA mineralocorticoid receptor antagonist SGLT2i sodium-glucose cotransporter-2 inhibitor

#### 2 Introduction

The TELEhealth and Dashboard Activated Health Services outreach (TELE-DASH) study is a pragmatic randomized controlled trial of a quality improvement (QI) intervention of a prospective panel management intervention to optimize medical treatment for Veterans with heart failure with reduced ejection fraction (HFrEF) compared to the receipt of usual VA health care services over a 6-month period of observation. The study will incorporate the existing VA Academic Detailing Heart Failure Dashboard (ADHFD) to target actionable patients with gaps in performance measures for guideline-directed medical therapies (GDMT). Patients with HFrEF are optimally managed by cardiovascular specialty clinics. Typically, patients are referred to cardiology or heart failure (HF) clinics from primary care, emergency department, or post-hospitalization clinicians and scheduled into clinic grids. These patients may be lost to follow-up, not referred without prior HF hospitalization, or clinicians may miss opportunities to optimize GDMT for HFrEF. GDMT includes Class I indicated medications from the following classes: beta blockers (BB), angiotensin-converting enzyme inhibitor (ACE), angiotensin II receptor blockers (ARB), angiotensin receptor neprilysin inhibitor (ARNI), mineralocorticoid receptor antagonist (MRA), sodium-glucose cotransporter-2 inhibitor (SGLT2i). <sup>1-3</sup> The intervention is designed around prospective panel management clinics led by clinicians using impromptu patient telephone calls or electronic communications with existing responsible clinicians.

## 3 Study Objectives

The purpose of this study is to measure the effectiveness of proactive panel management clinics to optimize GDMT relative to usual care. The study will also evaluate secondary outcomes that signify improved outcomes such as reduced hospitalizations and mortality. The study will also evaluate clinician time per intervention relative to usual cardiology or HF clinic structure.

# 4 Study Methods

### 4.1 General Study Design and Plan

This is a <u>randomized</u>, <u>pragmatic QI study</u> designed to evaluate the effectiveness of proactive panel management to close gaps in evidence-based care for patients with HFrEF. We will use the VA's ADHFD to generate a list of actionable patients with HFrEF and left ventricular ejection fraction (LVEF) ≤ 35%. After identifying a cohort of HFrEF patients from the ADHFD, we will <u>randomize individual patients</u> on the actionable list to usual VA care or a novel proactive panel management clinic. Clinicians will be trained on how to use the dashboard information to identify opportunities for optimization based on detailed chart review. The proactive panel management intervention will use clinicians to perform an electronic chart review and call patients impromptu at their discretion to evaluate HFrEF management and opportunities to optimize GDMT. Each panel management clinic is staffed by a single cardiovascular clinician or trainee with cardiology (PI) supervision. All patients will receive chart review or telehealth notes brought to the attention of primary care and cardiology clinicians. Patients randomized to the intervention will only receive one chart review during a half-day panel management clinic with follow-up of any laboratory results or diagnostic tests as required and referral to HF or general cardiology clinic as deemed appropriate. The control arm consists of the usual delivery of health services with routine scheduled appointments for primary care or cardiology.

Outcomes will be assessed at 6-months from the last patient to receive the intervention. The study is powered to detect superiority of the intervention compared to usual care in optimizing GDMT for HFrEF. Treatment assignment is based on 1:1 randomization using fixed blocks (size=6) to assure an equivalent number of patients randomized to the intervention and usual care. Patients are randomized after a list of 300 actionable patients

are generated from the ADHFD. Study participant numbers will be assigned to the list of patients sorted by optimization scores in Excel. The supervising statistician (AA) will generate concealed randomization assignments by participant identification numbers. The randomization assignments will be merged with baseline study dataset and exported as password protected Excel and PDF documents. Study investigators will divide the intervention arm into lists of 10 to 15 per half-day clinic. Patients not receiving chart review or phone call attempts will be reassigned to future panel management clinics until all patients receive the intervention. Patients that did not answer phone calls will receive chart review notes for primary care and cardiology clinicians and not be reassigned to future panel management clinics.

Study participants do not require informed consent as determined by the VA IRB review. Patients will receive all accepted standards of care and medications approved by the Food and Drug Administration for HFrEF indications. The VA Subcommittee for Research and Safety found an absence of any declared research-laboratory-based biohazards and granted exemption from continued review. The study will evaluate the effectiveness of the QI intervention, telephone/telemedicine panel management clinics, to more rapidly implement evidence-based care for patients with HFrEF. Patients in the usual care arm will be unaware they are part of the control group for the RCT. Intervention patients nor study staff are blinded to usual care or intervention assignments. Patients that receive the intervention will be informed this is a pilot quality improvement effort with informal consent before proceeding to the clinical interventions. Intervention patients may refuse to participate after being contacted by phone in the intervention.

Study enrollment is based on the inclusion and exclusion criteria used to filter the ADHFD list. A list of actionable patients with HFrEF will be exported for randomization. The GDMT optimization score will be automated for each patient on the extracted list (**Table 1**). A sample of 300 patients will be selected with the lowest GDMT composite scores. Once the final sample of the study is determined, patients will be randomized to usual care or the intervention. Intervention patients will be divided into smaller lists of 10 to 15 patients. These smaller lists will be assigned to proactive panel management clinics. Clinicians staffing the intervention clinics will review ADHFD data, review the electronic health record (EHR) and decide whether to proceed to evaluate and recommend treatment over the phone to patients directly. If clinicians did not have sufficient time to review all patients on their clinic list, they will be redistributed to future intervention clinics. Intervention clinics will be held until each patient assigned the intervention has a chart review or attempted telephone contact. A failure to contact a patient will trigger a letter to a patient or electronic communication to their primary care or cardiology clinician.

Prior to each ADHFD telehealth clinic (half-day clinic lasting 4 to 4.5 hours), clinicians will be sent a secure email that will include a password-protected Excel document of 15 patients with exported clinical summary data from the ADHFD. Clinicians will be instructed to chart-review patients and decide if an opportunity exists to further optimize the receipt of GDMT. Clinicians will also be given a document providing guidance on the sequence of GDMT optimization based on latest guidelines and VA policies (Supplement S1 GDMT Guidance Document). If a patient does not qualify for further optimization (i.e. chart documentation of prior intolerance, patient preference), a short note in the electronic health record (EHR) will document the chart review and inform the primary care clinician that based on chart review, no opportunity currently exists but they may consider further GDMT titration in the future. If a patient appears to have an opportunity for further titration, the clinician is encouraged to call the patient to see if they are available to discuss their HF care. If the patient agrees, a telehealth visit will take place over phone or switch to video. A formal telehealth cardiology visit will occur at the time of care. If the patient is interested but does not have time for a visit, a brief telephone note will be placed and a request for a future cardiology clinic visit will be requested. If a formal telehealth visit occurs, clinicians will be asked to inquire about key details around medication titration (Supplement S2 Interview

**Guide**). The data from chart review and interviews will be documented on a password-protected Excel document (**Supplement S3** Clinician Documentation Form). Any medication addition or titration will have indicated laboratory labs ordered per usual care. Lastly, clinicians will also be asked to administer a short survey with each participant based on a template at the end of the call proactive phone call (**Supplement S2 Interview guide**). Primary care and regular cardiology clinicians will be notified of any changes in medication management in the EHR. The study's lead (BZ, AV) will be available by phone to answer questions or problems that arise during the clinic. Supervision of patient encounters by clinical pharmacists, medical trainees, or advanced practice nurse practitioners and study protocols will be BZ as the licensed and boarded general cardiologist.

## 4.2 Inclusion-Exclusion Criteria and General Study Population

This quality improvement (QI) initiative involves patients with heart failure with reduced ejection fraction (HFrEF) receiving care in the VA West Los Angeles (WLA). The criteria for eligible patients are:

#### **Inclusion criteria:**

- Facility: Greater Los Angeles, CA
- Division: All divisions within Greater Los Angeles
- Patient is eighteen years of age or older
- Patients has a primary diagnosis of HFrEF (last documented LVEF ≤35% per ADHFD algorithms)
- Patient has an estimated GFR greater than or equal to 30 mL/min
- Patient lacks at least one active prescription of a beta-blocker, ACE/ARB/ARNI, MRA, or SGLT2i
- There are no cardiology appointments in the upcoming 2 weeks.

### **Exclusion criteria:**

Patient is currently hospitalized at WLA

# 4.3 Randomization and Blinding

Patients will be randomized 1:1 to intervention and usual care groups with all patients randomized at one time; given the target sample size of n=300 total patients, the sequence will be generated using permuted blocks of size 6 to ensure that an equal number of patients are randomized to panel management and usual care, maximizing efficiency (power). The randomization sequence will be concealed from the clinicians until after randomization has already been complete. Post-randomization, study staff will not be blinded to allocation. GLA IRB exemption was granted for consent of the low risk, non-experimental intervention. The intervention does not allow for blinding of participants in the intervention arm.

Figure 1: CONSORT Study Flow Diagram Template



# 5 Safety

Clinicians involved with the intervention will report acute kidney injury (AKI) defined as 25% decrease in GFR from baseline on follow-up labs (1-week for MRA and 1-2 weeks for ACE/ARB/ARNI) after a successful medication titration within the intervention group. Laboratory alerts will be followed by pilot study clinicians. Hospitalization related to adverse medication event (e.g. symptomatic hypotension, AKI, hyperkalemia) related to the intervention. Difference in mortality between intervention and usual care.

#### 6 Adverse Events

Specific adverse events of interest include symptomatic hypotension documented in the EHR. Hospitalizations related to heart failure will be captured during the study end using the ADHFD. If patients were removed from the dashboard at 6 months, a chart review will be performed to abstract missing data.

## 7 References

- 1. McMurray JJV, Solomon SD, Inzucchi SE, et al. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. *N Engl J Med*. 2019;381(21):1995-2008. doi:10.1056/nejmoa1911303
- 2. Packer M, Anker SD, Butler J, et al. Cardiovascular and Renal Outcomes with Empagliflozin in Heart Failure. *N Engl J Med*. 2020;383(15):1413-1424. doi:10.1056/nejmoa2022190
- 3. Maddox TM, Januzzi JL, Allen LA, et al. 2021 Update to the 2017 ACC Expert Consensus Decision Pathway for Optimization of Heart Failure Treatment: Answers to 10 Pivotal Issues About Heart Failure With Reduced Ejection Fraction: A Report of the American College of Cardiology Solution Set Oversig. *J Am Coll Cardiol*. 2021;77(6):772-810. doi:10.1016/j.jacc.2020.11.022

# 8 Listing of Tables, Listings, and Figures

Figure 1: CONSORT Study Flow Diagram Template

8

## 9 Supplemental Material

#### S1: GDMT Guidance Document for LVEF ≤35%

#### I. Make a recommendation

Step 1: patient not at target ACE/ARB or beta-blocker

Initiate/titrate up ACE/ARB and/or beta blocker

- If signs of volume overload or HR<70 → ACE/ARB
- If signs of euvolemia, HR>70, atrial fibrillation history, ventricular ectopy → Beta-blocker
- Age < 75, systolic BP>120 mm Hg, HR >70, normal renal function → Start both

## Tailored based on patient's profile and history.

Step 2a: Transition ACE/ARB to ARNI

- Initiate ARNI once patient is taking equivalent dosing to lisinopril 20 mg daily

Step 2b: Initiate and titrate up aldosterone antagonist

- If K < 5 (helpful for hypokalemia)</li>
- Well tolerated in low BP patients
- Check labs 3-7 days within initiation. Repeat labs monthly for the first 3 months.

## Step 2c:

Initiate SGLT2i – empagliflozin 10mg daily

- Initiate earlier if A1C ≥7% or GFR 25-60 mL/min/1.73m<sup>2</sup> refer nephrology for SGLT2i
- Otherwise, add to cornerstone beta-blocker and RAAS inhibitor, ideally when dosing is stable.

## II. Discuss instructions and precautions

Symptomatic hypotension, genital yeast infections (SGLT2i)

#### III. Recommended follow-up

Labs, diagnostic imaging or studies, new consults, follow-up appointments

### Strategies for intolerance/symptomatic hypotension

- Reduce non-GDMT antihypertensives, half diuretic dose with initiation of RAAS inhibitor or SGLT2i.
- Consider insulin reduction for history hypoglycemic events with SGLT2i.
- Space out administration times for medications
- Move RAAS inhibitors to evening to peak during sleep
- Lower morning doses relative to evening doses



#### **S2: Interview Guide**

| In | ۲r | വ | ดเ | Ш | CŤ | ın | n |
|----|----|---|----|---|----|----|---|

Hello, I am Dr. \_\_\_\_\_ calling from the West LA VA Cardiology. We are piloting an effort to proactively reach out to Veterans with heart disease to see how they are doing and improve their medical therapies for heart failure. Is now a convenient time to discuss your heart medications?

- Yes: Thank you. Do you have access to a smartphone or computer? May we convert this visit to video?
- No: May we request a follow-up phone, video, or in-person visit with our heart failure clinic?

Yes: Thank you. [RTC WLA-Cardiomyopathy Clinic]

**No:** Thank you for your time. [Chart review note for PMD and last cardiology fellow/attending highlighting potential opportunity for further medication optimization]

# Obtain history and assess functional NYHA class

- 1. How have you been feeling? Any change in [dyspnea/orthopnea/edema]?
- 2. What type of physical activities do you do regularly [walking, exercise, stairs]?
- 3. Do you know what medications you take for heart failure and how do manage your medications?
- 4. Have you had issues with any of heart failure medications in the past?
- 5. Do you check your home blood pressure and weights regularly? What are they?
- 6. Do you have issues with lightheadedness/dizziness or passing out?

| Make recommendatio | n |
|--------------------|---|
|--------------------|---|

| Optimization: I see that you might benefit from an increase in yo | ou/ I see that you might benefit from an |
|---|---|
| additional medication/I see you may benefit from stoppi | ng one of your non-heart failure blood |
| pressure medications. May we start that today and you can rece | ive the medication in the mail or pick-up from |
| your local VA clinic? | |

Hypervolemia: Increase diuretic regimen and refer for face to face visit within 1 week.

## <u>Discuss appropriate precautions with optimization</u>

Dizziness, orthostasis, follow-up blood tests. SGLT2i [genital yeast infections/hypoglycemia for IDDM]

## Next steps

- Order medications
- Follow-up appointment
- Required labs
- BMP in one week (MRA), 1-2 weeks (ACE/ARB/ARNI)

#### Questions

Do you have any concerns related to medication change? Other questions?

#### Feedback

Thank you for your time. This was a call part of our pilot telephone heart clinic program. How would you rate your experience with the heart failure outreach today on a scale 1 to 10 (10 being very appreciated)? Any suggestions to improve the program?

# **S3: Clinician Documentation Form**

Documentation survey which will guide clinician's chart review and patient conversation. The form will be password-protected and utilize checkbox and short answers for clinician ease.

| Clinic | Clinician | Start | Homeless | Active | Female | Last | Last cards | Last PCP appt |
|---|---|---|---|---|---|---|---|---|
| Date | | Time | | Substance Use | | EF | appt | |
| 1/1/21 | Ziaeian, | 13:55 | х | х | Х | 35- | 1/1/21 | 1/1/21 |
| | Boback | | | | | 40% | | |

| Phone Call Time | NYHA Class | No Response |
|-----------------|------------|-------------|
| 9 minutes | III | Х |

| Reasons for no GDMT titration | | | | |
|---|---|---|---|---|
| Prior intolerance Prior adverse event Patient declined Patient concerned of side effects Other | | | | |
| Х | Х | Х | х | Cost |

| Actions Performed | | | | | | |
|---|---|---|---|---|---|---|
| Number of Rx adjusted | Med adjustment | Labs<br>ordered | Imaging / diagnostic tests | RTC | Patient Letter | Consults |
| 3 | Amlodipine stopped | х | Х | х | х | Х |

| Feedback | End Time | Comments |
|----------|----------|-----------------------|
| 9 | 1415 | Straight to voicemail |

| <b>Clinician Documentation</b> | form definitions |
|---|---|
| Clinic date | Date today, (mm/dd/yy) |
| Clinician | Name of clinician (Last, First) |
| Start Time | Military time at onset of pre-chart |
| Homeless | Is the veteran currently experiencing homelessness? |
| Active substance use | Is the veteran actively using substances? |
| Female | Sex as categorized in EHR |
| Last EF | Most recent left ventricular ejection fraction on transthoracic echocardiogram, % |
| Last cards appt | Date of last cardiology clinic visit, (mm/dd/yy) |
| Last PCP appt | Date of last PCP visit, (mm/dd/yy) |
| Phone Call Time | Duration of successful phone or video visit |
| NYHA Class | Based on patient's symptoms and chart review, (1-3) |
| No response | Indication if no response after 2 attempts |
| Patient requests later appointment | Indication if patient is interested in further discussion, but busy at this time. Check and order RTC cardiology |
| Reasons for no GDMT | |
| Prior intolerance | History of symptomatic bradycardia or hypotension on GDMT |
| Prior adverse event | History of hospitalization or angioedema related to GDMT titration. History of yeast infection while taking an SGLT2i inhibitor |
| Patient declined | Patient declined additional or higher doses of medications in the past |
| Patient concerned of side | |
| effects | Patient is concerned of side effects of GDMT |
| Other | Other reasons cited by patients or on chart review in the comments |
| Actions Performed | |
| # medication adjustments | Number of medications adjusted after this visit |
| Medication adjustment detail | Description of medication adjustment |
| Labs ordered | If laboratory tests ordered as part of today's plan |
| Imaging / diagnostic tests ordered | If imaging or diagnostic tests ordered as part of today's plan |
| RTC | If "return to clinic" order placed to patient's cardiology clinic |
| Patient Letter | Letter mailed to patient regarding following up with primary care or cardiology regarding heart failure. |
| New consults | If new consults placed as part of today's plan |
| Patient feedback | Self-reported experience of conversation and heart failure plan, on a scale of 1 to 10, where 1 means an awful experience and 10 means an exceptional experience |
| Time (end call) | Military time on completion of phone call |
| Comments | Noteworthy general observations not contained in fields regarding chart review or patient experience |